CLINICAL TRIAL: NCT02234934
Title: A Two-Part, Phase I/II, Non Randomized, Multicenter, Open-Label Study of G1XCGD (Lentiviral Vector Transduced CD34+ Cells) in Patients With X-Linked Chronic Granulomatous Disease
Brief Title: Study of Gene Therapy Using a Lentiviral Vector to Treat X-linked Chronic Granulomatous Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Boston Children's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Genethon (Other); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Donald B. Kohn, M.D., Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G1XCGD; 2P01HL073104 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Granulomatous Disease, Chronic, X-linked
Keywords: Gene Therapy; X-Linked Chronic Granulomatous Disease (X-CGD); Lentiviral Vector
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lentiviral G1XCGD Gene Therapy, Part A (Experimental): Transplantation with autologous CD34+ stem cells corrected with X1XCGD lentiviral vector after myeloreductive conditioning
  Interventions: Biological: Lentiviral G1XCGD Gene Therapy
- Lentiviral G1XCGD Gene Therapy, Part B (Experimental): Transplantation with autologous CD34+ stem cells corrected with X1XCGD lentiviral vector after modified myeloreductive conditioning including increased monitoring and rescue treatment
  Interventions: Biological: Lentiviral G1XCGD Gene Therapy

INTERVENTIONS:
Biological: Lentiviral G1XCGD Gene Therapy — The investigational product is patient-specific and corresponds to autologous CD34+ cells transduced ex vivo with the G1XCGD vector in their final suspension. The starting materials used for the production of the investigational product consist of the viral vector and the patient's CD34+ cells.
  The G1XCGD vector is used to transduce autologous CD34+ cells ex vivo. These transduced cells are then frozen, and an aliquot tested and characterized for quality. If the cell product passes release criteria, it is thawed at bedside and infused into the patient after the patient has received myelo-ablative conditioning. The cell/product dose will consist of at least 3 x 10^6 cells per kg of body weight transduced ex vivo with 1 x 10^8 IG/mL of lentiviral vector to achieve > 0.3 integrated copies per cell.
  Other Names: G1XCGD (pCCLChimGp91/VSVg lentiviral vector)

SUMMARY:
Chronic Granulomatous Disease (CGD) is an inherited immunodeficiency disorder which results from defects that prevent white blood cells from effectively killing bacteria, fungi and other microorganisms. Chronic granulomatous inflammation may compromise vital organs and account for additional morbidity. CGD is thought to affect approximately 1 in 200,000 persons, although the real incidence might be higher due to under-diagnosis of milder phenotypes.

The first gene therapy approaches in X-CGD have shown that effective gene therapy requires bone-marrow (BM) conditioning with chemotherapy to make space for the gene-modified cells to engraft. These studies demonstrated that transplantation of gene modified stem cells led to production of white blood cells that could clear existing infections. However, some trials using mouse-derived retroviral vectors were complicated by the development of myelodysplasia and leukemia-like growth of blood cells. This trial will evaluate a new lentiviral vector that may be able to correct the defect, but have much lower risk for the complication.

This study is a two-part, prospective non-controlled, non-randomized Phase I/II clinical trial to assess the safety, feasibility and efficacy of cellular gene therapy in patients with chronic granulomatous disease using transplantation of autologous bone marrow CD34+ cells transduced ex vivo by the G1XCGD lentiviral vector containing the human CGD gene. Primary objectives include evaluation of safety and evaluation of efficacy by biochemical and functional reconstitution in progeny of engrafted cells and stability at 12 months. Secondary objectives include evaluation of clinical efficacy, longitudinal evaluation of clinical effect in terms of augmented immunity against bacterial and fungal infection, transduction of CD34+ hematopoietic cells from X-CGD patients by ex vivo lentivirus-mediated gene transfer, and evaluation of engraftment kinetics and stability. Approximately 3-6 patients will be treated per site with a goal of 16 total patients to be treated with G1XCGD lentiviral vector.

DETAILED DESCRIPTION:
The therapeutic product to be evaluated is autologous CD34+ hematopoietic stem cells (HSC) modified by ex vivo transduction using the pCCLchimGP91WPRE lentiviral vector (G1XCGD Modified Autologous BM CD34 cells) containing the human CGD gene. The G1XCGD lentiviral vector is a 3rd generation self-inactivating lentiviral vector which directs gp91phox expression from a codon-optimized form of the CYBB gene preferentially to myeloid cells, with a modified WPRE (PRE4).

G1XCGD is an integrative, 3rd generation replication-defective, self-inactivating (SIN) HIV-derived Lentiviral (LV) vector, with a mutated Woodchuck hepatitis virus Posttranscriptional Regulatory Element (WPRE) sequence. A LV vector derived from HIV-1 has been chosen with respect to LV natural properties: they are genetically stable, permanently integrate into the genome of transduced cells and provide long-term gene expression in vitro and in vivo. The transduction of Hematopoietic Stem Cells (HSC) with such LV can be achieved after limited pre-activation of the cells in short-term cultures with cytokines, in conditions that are compatible with the preservation of the self-renewing capacities of these cells. These properties make these LV suitable for ex-vivo gene therapy strategies using HSC.

G1XCGD provirus includes a chimeric promoter designed to regulate the transgene expression in myeloid cells and a transgene called GP91 (also known as CYBB), which is a codon-optimized cDNA sequence of the human CYBB gene also known as GP91-PHOX or NOX2 gene. The promoter is a synthetic chimeric element created by the fusion of c-Fes and Cathepsin G minimal 5'-flanking regions. Cathepsin G is a serine protease stored in the azurophil granules of neutrophil granulocytes. Part of the chimeric promoter contains binding sites for myeloid transcription factors C/EBP and PU.1 from the upstream region of the transcription start site of the Cathepsin G gene. The other part of the chimeric promoter is a human c-Fes sequence that has been added to enhance the Cathepsin G promoter activity in granulocytic cells. The resulting chimeric promoter is able to i) regulate the expression of the GP91 transgene in myeloid cells in a specific manner, and ii) to effectively restore NADPH-oxidase activity in granulocytes, as reported by Santilli et al. (Santilli et al., 2011) and confirmed in preclinical studies conducted with the G1XCGD vector. The GP91 transgene codes for the 570 amino-acid cytochrome b-245, a 91 kD beta polypeptide that is also known as the NADPH-oxidase catalytic subunit gp91-phox, or cytochrome b-245 heavy chain, or gp91-phox protein.

ELIGIBILITY:
Inclusion Criteria:

(Part A & B)

* Male X-CGD patients > 23 months of age
* Molecular diagnosis confirmed by DNA sequencing and supported by laboratory evidence for absent or reduction > 95% of the biochemical activity of the NADPH-oxidase
* At least one prior, ongoing or refractory severe infection and/or inflammatory complications requiring hospitalization despite conventional therapy
* No 10/10 HLA-matched donor available after initial search of NMDP registries
* No co-infection with Human Immunodeficiency Virus (HIV)-1 or -2, hepatitis B virus or hepatitis C virus, adenovirus, parvovirus B 19 or toxoplasmosis, or active infection with CMV
* Written informed consent for adult patient, and assent for pediatric subjects seven years or older.
* Parental/guardian and, where appropriate, child's signed consent/assent

Exclusion Criteria:

* Age < 23 months
* 10/10 HLA identical (A,B,C,DR,DQ) family or unrelated or cord blood donor unless there is deemed to be an unacceptable risk associated with an allogeneic procedure
* Contraindication for leukapheresis or bone marrow harvest (anemia Hb <8g/dl, cardiovascular instability, severe coagulopathy)
* Appropriate organ function as outlined below must be observed within 8 weeks of entering this trial.

  1. Hematologic

     1. Anemia (hemoglobin < 8 g/dL).
     2. Neutropenia (absolute granulocyte count <1,000/mm3)
     3. Thrombocytopenia (platelet count < 150,000/mm3).
     4. PT or PTT > 2X the upper limits of normal (patients with a correctable deficiency controlled on medication will not be excluded).
     5. Cytogenetic abnormalities known to be associated with hematopoietic defect on peripheral blood or bone marrow.
  2. Infectious

     a. Evidence of co-infection with HIV-1, HIV-2, hepatitis B, Hepatitis C, adenovirus, parvovirus B19, toxoplasmosis. CMV infection is allowable as long as the infection is under control.
  3. Pulmonary

     a. Resting O2 saturation by pulse oximetry < 90% on room air.
  4. Cardiac

     1. Abnormal electrocardiogram (EKG) indicating cardiac pathology.
     2. Uncorrected congenital cardiac malformation with clinical symptomatology.
     3. Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension.
     4. Poor cardiac function as evidenced by LV ejection fraction < 40% on echocardiogram.
  5. Neurologic

     1. Significant neurologic abnormality by examination.
     2. Uncontrolled seizure disorder.
  6. Renal

     1. Renal insufficiency: serum creatinine ≥ 1.5 mg/dl, or ≥ 3+ proteinuria.
     2. Abnormal serum sodium, potassium, calcium, magnesium, phosphate at grade III or IV by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  7. Hepatic/GI:

     1. Serum transaminases > 5X the upper limit of normal (ULN).
     2. Serum bilirubin > 2X ULN.
     3. Serum glucose > 1.5x ULN.
  8. Oncologic

     a. Evidence of active malignant disease
  9. General

     1. Expected survival < 6 months
     2. Major congenital anomaly
     3. Ineligible for autologous HSCT by the criteria at the clinical site.
     4. Contraindication for administration of conditioning medication. (Known sensitivity to Busulfan)
     5. Administration of gamma-interferon within 30 days before the infusion of transduced, autologous CD34+ cells.
     6. Participation in another experimental therapeutic protocol within 6 months prior to baseline and during the study period.
     7. Tested positive (definitive) for the presence of multiple types (2 or more) of anti-platelet antibodies.
     8. Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful study completion.
     9. Patient/Parent/Guardian unable or unwilling to comply with the protocol requirements.

Part B Additional exclusion criteria:

* Patients >12 years of age at enrolment
* Patients ≤12 years of age with a body weight >40kg at enrolment

Min Age: 23 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events assessed by CTCAE v4 | up to 2 years
  Record clinical significant adverse events, laboratory abnormalities, monitor overall adverse events for the study as a whole, including serious adverse events
Measuring percentage of subjects who have ≥ 10% oxidase positive granulocytes | At month 12 after transplant
  Oxidase positive granulocytes for each subject will be assessed by DHR flow cytometry

OTHER OUTCOMES:
Concentration of gp91 protein produced in response to the corrected gene | up to 2 years
  We will look for the presence of gp91 antibodies in blood
Characterization of drug product immunophenotype | up to 2 years
  Different lymphocyte subsets using flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Donald B. Kohn, MD, Study Chair — University of California, Los Angeles; Caroline Y. Kuo, MD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - National Institutes of Health, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Results will be published in scientific literature once trial is completed and data analysis is done.

REFERENCES:
- [Background] Santilli G, Almarza E, Brendel C, Choi U, Beilin C, Blundell MP, Haria S, Parsley KL, Kinnon C, Malech HL, Bueren JA, Grez M, Thrasher AJ. Biochemical correction of X-CGD by a novel chimeric promoter regulating high levels of transgene expression in myeloid cells. Mol Ther. 2011 Jan;19(1):122-32. doi: 10.1038/mt.2010.226. Epub 2010 Oct 26. PMID 20978475
- [Derived] Brendel C, Rothe M, Santilli G, Charrier S, Stein S, Kunkel H, Abriss D, Muller-Kuller U, Gaspar B, Modlich U, Galy A, Schambach A, Thrasher AJ, Grez M. Non-Clinical Efficacy and Safety Studies on G1XCGD, a Lentiviral Vector for Ex Vivo Gene Therapy of X-Linked Chronic Granulomatous Disease. Hum Gene Ther Clin Dev. 2018 Jun;29(2):69-79. doi: 10.1089/humc.2017.245. Epub 2018 Apr 17. PMID 29664709